CLINICAL TRIAL: NCT06538688
Title: Evaluation of Orthodontic Extrusion of Impacted Mandibular Third Molar in Close Proximity to Inferior Alveolar Nerve Prior to Extraction ( a Clinical Trial)
Brief Title: Orthodontic Extrusion of High Risk Impacted Mandibular Third Molar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Azza Mohamed Elmetwally Elmetwally, Dentist, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OEIMTM
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Inferior Alveolar Nerve Injuries
Keywords: Orthodontic extraction; impacted third molar; TAD
MeSH Terms: conditions — Mandibular Nerve Injuries

STUDY DESIGN:
Intervention Model Description: Patients with impacted mandibular third molar in close proximity to the inferior alveolar nerve requiring orthodontic extrusion of the impacted teeth before extraction
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Patients with impacted mandibular third molar in close proximity to the inferior alveolar nerve
  Interventions: Procedure: Orthodontic extrusion of the impacted mandibular third molar by using the maxillary miniscrew and cross arch elastic power chain as a temporary anchorage device before extraction

INTERVENTIONS:
Procedure: Orthodontic extrusion of the impacted mandibular third molar by using the maxillary miniscrew and cross arch elastic power chain as a temporary anchorage device before extraction — Orthodontic extrusion of the impacted mandibular third molar of high-risk for nerve injury using maxillary TAD.
  Other Names: Using temporary anchorage device (TAD)in the maxillary bone for traction of the impacted tooth before extraction

SUMMARY:
The goal of this clinical trial is to investigate the usage of maxillary miniscrew and cross-arch elastics for the orthodontic traction of the impacted mandibular third molar in close proximity to the inferior alveolar nerve to decrease the chance of nerve injury

DETAILED DESCRIPTION:
To investigate the traction of the impacted mandibular third molar away from the inferior alveolar nerve by using the orthodontic miniscrew in the maxillary bone and cross-arch elastic power chain as a temporary anchorage device before extraction to avoid injury of the nerve and neurosensory complications.

ELIGIBILITY:
Inclusion Criteria:

* patients with impacted mandibular third molar in close proximity to the inferior alveolar nerve.
* Cooperative patients free of chronic diseases which interfere with needed results (e.g.diseases affect the bone regeneration ).
* Patients with good oral hygiene.

Exclusion Criteria:

* patients with limitation in mouth opening.
* patients with mental or physical disabilities.
* Allergy to anaesthetic components or antibiotics.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2023-12-17 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Radiographically | 6months
  By measuring the amount of extrusion of the impacted tooth gained in millimetres Using CBCT

SECONDARY OUTCOMES:
Clinical neurosensory assessment | 6months
  By using pinprick test in which ;A sharp dental probe was applied to the skin over chin region, lip and mucosa in a quick pricking movement and pain perception of the patient was assessed. Each area was tested three times bilaterally.the scale ranged from 0-2, where 0= no sensation, 1= decreased sensation and 2= normal sensation.
clinical brush stroke directional test | 6months
  using a micro brush tip which was moved in horizontal and/or vertical directions on the chin area ten times and asked the patient to reproduce the movements the scale ranged from 0-2, where 0= no sensation, 1= decreased sensation and 2= normal sensation.
Clinical Two-point discrimination test | 6months
  By using probes of caliper device which were drawn across the skin at constant pressure and patient was asked whether one or two points were felt, the minimum separation distance was felt by the patient was termed two point discrimination threshold.scoring from 0-2 in which; 0=>15mm, 1=8-15, 2= <8 .

CONTACTS AND LOCATIONS:
Overall Officials: Saeeda Osman, Professor Dr, Study Chair — Alexandria University; Tarek Nasreldin, Ass.prof., Study Director — Alexandria University; Tasneem Amer, Lecturer, Study Director — Alexandria University
Locations (3):
- Egypt (3):
  - Alexandria university, Alexandria
  - Faculty of Dentistry, Alexandria University, Alexandria
  - Faculty of Dentistry, Alexandria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jung S, Lee JH, Huh J, Park W. Orthodontic Extrusion of Mandibular Third Molar With a Miniscrew and Cross-Arch Elastic. J Oral Maxillofac Surg. 2021 Jul;79(7):1422.e1-1422.e8. doi: 10.1016/j.joms.2021.01.036. Epub 2021 Feb 7. PMID 33667345
- [Background] Kim JW, Cha IH, Kim SJ, Kim MR. Which risk factors are associated with neurosensory deficits of inferior alveolar nerve after mandibular third molar extraction? J Oral Maxillofac Surg. 2012 Nov;70(11):2508-14. doi: 10.1016/j.joms.2012.06.004. Epub 2012 Aug 15. PMID 22901857
- [Background] Ramaraj PN. Orthodontic extraction: the riskless extraction of the impacted lower third molars close to the mandibular canal. J Oral Maxillofac Surg. 2008 Jun;66(6):1317; author reply 1317. doi: 10.1016/j.joms.2008.02.008. No abstract available. PMID 18486807
- [Background] Kalantar Motamedi MR, Heidarpour M, Siadat S, Kalantar Motamedi A, Bahreman AA. Orthodontic Extraction of High-Risk Impacted Mandibular Third Molars in Close Proximity to the Mandibular Canal: A Systematic Review. J Oral Maxillofac Surg. 2015 Sep;73(9):1672-85. doi: 10.1016/j.joms.2015.03.031. Epub 2015 Mar 24. PMID 25882437
- [Background] Alessandri Bonetti G, Bendandi M, Laino L, Checchi V, Checchi L. Orthodontic extraction: riskless extraction of impacted lower third molars close to the mandibular canal. J Oral Maxillofac Surg. 2007 Dec;65(12):2580-6. doi: 10.1016/j.joms.2007.06.686. No abstract available. PMID 18022488
- [Result] Zhao S, Wang Y, Yang X, Zhou X, Wang Z, Zhang K, Yang X. Extraction of impacted mandibular third molars in close proximity to the inferior alveolar canal with coronectomy-miniscrew traction to avoid nerve injury. Clin Oral Investig. 2023 Aug;27(8):4279-4288. doi: 10.1007/s00784-023-05044-9. Epub 2023 Jun 16. PMID 37326659